CLINICAL TRIAL: NCT04866095
Title: Inferior Vena Cava Compliance in Trans-thoracic Echocardiography: is the Trans-hepatic Window as Reliable as the Subcostal One
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of anesthesiology department, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-WICAVE
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Surgical Procedure, Unspecified
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery (Experimental): All patients, who have given their consent, aged over 18 years, with a sinus rhythm, requiring a surgical procedure that allows obtaining high quality transthoracic echocardiogram imaging without pain and discomfort.
  Interventions: Device: Transthoracic echocardiogram; Device: Clear Sight system

INTERVENTIONS:
Device: Transthoracic echocardiogram — Transthoracic echocardiogram (TTE) is a widely used and validated imaging technique which involves the study of the heart and great vessels through multiple examination windows. In particular, the subcostal window represents the gold standard for evaluating the diameter of the inferior vena cava (IVC) and its compliance, allowing the physician to obtain valuable information on the volume status of patients. Acquiring images in the subcostal window with a transthoracic echocardiogram (TTE) can be, in some cases, difficult or impossible due to the presence of drainages or surgical wounds: in such cases an alternative could be represented by the trans-hepatic window. This has not been validated in the scientific litterature.
Device: Clear Sight system — The Clear Sight System is a non-invasive blood pressure (BP) monitoring system, where the CO is determined analysing the photo-plethysmography curve by a miniaturized pressure cuff and infrared LEDs.
  Its main advantage is to assess CO continuously in a completely non-invasive way, following its variations and thereby contributing to the detection of hypovolaemia. Other visualized parameters are: the stroke volume (SV), the systemic vascular resistance (SVR) as well as the BP and the heart rate (HR).

SUMMARY:
The ability to assess intravascular volume is an essential part of perioperative care: insufficient intravascular volume can result in decreased oxygen delivery to tissues and organ dysfunction, while fluid overload can contribute to the development of oedema, organ dysfunction, respiratory failure and healing defect.

At the present state, there are many different methods of interpreting intravascular circulating blood volume. Non-invasive techniques such as the Clear Sight System, and the transthoracic echocardiogram (TTE) have been proposed as non-invasive methods to assess patient' blood volume.

The aim of this study is to assess whether the measure of the inferior vena cava (IVC) in the trans-hepatic window is as reliable as in the subcostal window to determine fluid responsiveness in perioperative patients. In this study, preload increase will be obtained through passive leg raising. Sensibility and specificity of the two echocardiographic approaches to predict fluid responsiveness will be compared while using the subcostal window as the "gold standard". The effect of passive leg elevation on patient's cardiac output response will be assessed with two different non-invasive techniques: the Clear Sight system and the TTE.

DETAILED DESCRIPTION:
The ability to assess intravascular volume is an essential part of perioperative care: insufficient intravascular volume can result in decreased oxygen delivery to tissues and organ dysfunction, while fluid overload can contribute to the development of oedema, organ dysfunction, respiratory failure and healing defect.

Assessment of the volume status in perioperative patients relies on two important concepts: euvolemia and fluid responsiveness.

Euvolemia describes a state of adequate circulating blood volume that allows suitable filling of the cardiac chambers making possible for the heart to produce a cardiac output that meets the peripheral oxygen demand.

Fluid responsiveness describes the ability of the heart to adapt blood flow in response to preload increase.

As euvolemia is the ultimate goal of fluid administration then evaluating fluid responsiveness reflects the process of working toward establishing euvolemia.

At the present state, there are many different methods of interpreting intravascular circulating blood volume: those related to pressures measurements: the central venous pressure (CVP), the pulmonary artery occluded pressure (PAOP), and those related to cardiac output measurements like thermodilution and pulse contour techniques. It is worth noting that all these are invasive methods that expose patients to a series of possible side effects such as: pneumothorax, infections, hematomas and vascular lesions. Non-invasive techniques such as the Clear Sight System, and the transthoracic echocardiogram (TTE) have been proposed as non-invasive methods to assess patient' blood volume.

TTE is a widely used and validated imaging technique which involves the study of the heart and great vessels through multiple examination windows.

In particular, the subcostal window represents the gold standard for evaluating the diameter of the inferior vena cava (IVC) and its compliance, allowing the physician to obtain valuable information on the volume status of patients: several studies have reported that these measurements could predict accurately the hemodynamic response of patient to a change in cardiac preload. However, acquiring images in the subcostal window can be, in some cases, difficult or impossible due to the presence of drainages or surgical wounds; in such cases an alternative could be represented by the trans-hepatic window which, at the best of the investigator's knowledge, it has never been validated in the literature.

The Clear Sight System is a non-invasive blood pressure (BP) monitoring system, where the CO is determined analysing the photo-plethysmography curve by a miniaturized pressure cuff and infrared LEDs.

Its main advantage is to assess CO continuously in a completely non-invasive way, following its variations and thereby contributing to the detection of hypovolaemia. Other visualized parameters are: the stroke volume (SV), the systemic vascular resistance (SVR) as well as the BP and the heart rate (HR).

Passive leg raising (PLR) is a test developed to predict patient's hemodynamic response to increase preload without any fluid administration. Raising the patient from a semi-recumbent position to a position with the head at 0° and the legs raised to a 45° angle is associated with about 300 ml of blood volume mobilization from the lower limbs and splanchnic territory to the central compartment resulting in increased venous return to the heart. This manoeuvre provokes a preload increase to which patients could respond with (responder) or without (non-responders) an augmentation of their cardiac output.

The aim of this study is to assess whether the measure of the IVC in the trans-hepatic window is as reliable as in the subcostal window to determine fluid responsiveness in perioperative patients. In this study, preload increase will be obtained through passive leg raising. Sensibility and specificity of the two echocardiographic approaches to predict fluid responsiveness will be compared while using the subcostal window as the "gold standard". The effect of passive leg elevation on patient's cardiac output response will be assessed with two different non-invasive techniques: the Clear Sight system and the TTE.

ELIGIBILITY:
Inclusion Criteria:

All patients of the CHU Brugmann hospital, who have given their consent, aged over 18 years, with a sinus rhythm, requiring a surgical procedure that allows obtaining high quality TTE imaging without pain and discomfort.

Examples of such surgeries are:

* Orthopaedic surgery: interventions of upper limbs.
* Stomatology: dental extractions
* Gastroenterology: oesophagus gastroscopy
* Maxillo-facial surgery: septoplasties, rhinoplasties, Le Fort surgeries
* ENT surgery: thyroidectomy, sleep endoscopies
* Gynaecology: hysteroscopy, voluntary terminations of pregnancy
* Ophthalmic surgery

Exclusion Criteria:

* Refusal to participate to the study
* suboptimal image acquisition
* atrial fibrillation, patients with 6 or more extra systoles per minute
* cardiac valvular pathologies
* TTE imaging causing pain and/or discomfort to the patient
* surgeries that don't allow obtaining high quality imaging, elevated intra-abdominal pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Difference of sensitivity between the trans-hepatic window versus the subcostal window with TTE | 20 minutes
  Comparison of the sensitivity of both the trans-hepatic window and the subcostal window to predict the cardiac output response by transthoracic echocardiogram (TTE) to passive leg raising.
Difference of specificity between the trans-hepatic window versus the subcostal window with TTE | 20 minutes
  Comparison of the specificity of both the trans-hepatic window and the subcostal window to predict the cardiac output response by transthoracic echocardiogram (TTE) to passive leg raising.

SECONDARY OUTCOMES:
Difference of sensitivity between the trans-hepatic window versus the subcostal window with the Clear Sight system | 20 minutes
  Comparison of the sensitivity and specificity of both the trans-hepatic window and the subcostal window to predict the cardiac output response (with the Clear Sight system) to passive leg raising.
Difference of specificity between the trans-hepatic window versus the subcostal window with the Clear Sight system | 20 minutes
  Comparison of the sensitivity and specificity of both the trans-hepatic window and the subcostal window to predict the cardiac output response (with the Clear Sight system) to passive leg raising.
Right atrial pressure (RA)- trans-hepatic window | 20 minutes
  Evaluation of the estimation of RA pressure obtained with the trans-hepatic and sub-costal approaches
Right atrial pressure (RA) - subcostal window | 20 minutes
  Evaluation of the estimation of RA pressure obtained with the trans-hepatic and sub-costal approaches
Cardiac output | 20 minutes
  Cardiac output calculated by: CO= sub-Aortic Velocity Time Integral (sAoVTI) × heart rate in beats per minute (bpm) × left ventricular outflow track (LVOT)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zuccarini, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No